CLINICAL TRIAL: NCT03283592
Title: Review and Assessment of Network Meta-analyses for Knowledge Uptake (RANK) Study
Brief Title: Review and Assessment of Network Meta-analyses for Knowledge Uptake Study
Acronym: RANK
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: did not receive funding to conduct study
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 17-0107
Record Dates: First submitted 2017-09-11; First posted 2017-09-14 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Clinical Decision-making

STUDY DESIGN:
Intervention Model Description: 2-arm, parallel assignment
Who Masked: Outcomes Assessor
Masking Description: Single blind (outcome assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rank-Heat Plot (Experimental): The intervention group will receive an online survey to evaluate their interpretation of the results from the NMA with a rank-heat plot including results from 2 outcomes that were selected by our knowledge users (#injurious falls, #fractures).
  Interventions: Other: Rank-Heat Plot
- SUCRA (surface under the cumulative ranking) Plot (Active Comparator): The control group will receive an online survey to evaluate their interpretation of the results from the NMA with the SUCRA plots including results from the same 2 outcomes that will be presented to the intervention group (i.e., #injurious falls, #fractures).
  Interventions: Other: SUCRA Plot

INTERVENTIONS:
Other: Rank-Heat Plot — provides a visual presentation of treatment hierarchy across multiple outcomes
  Arms: Rank-Heat Plot
Other: SUCRA Plot — provides a visual presentation of treatment ranking for a single outcome.
  Arms: SUCRA (surface under the cumulative ranking) Plot

SUMMARY:
This randomized controlled trial will assess the interpretability of the rank-heat plot for presenting the results of network meta-analysis in comparison to SUCRA (surface under the cumulative ranking) plots which are suggested to present one of the best ranking statistics.

DETAILED DESCRIPTION:
Clinicians are responsible for making decisions to improve health outcomes. When available, clinicians should use the results of a knowledge synthesis, such as systematic reviews and meta-analyses, to inform decision-making. Pairwise meta-analyses are limited, however, by the availability of RCTs that directly compare interventions. This is troublesome for knowledge users who require results from comparisons of multiple interventions to inform decision-making. To address this concern, the use of network meta-analyses (NMAs) is increasing in healthcare the literature. NMAs are a useful tool because they can summarize results from numerous studies and interventions. It is unclear how NMA results should be presented to increase the likelihood of clinicians understanding and using the results to improve health outcomes. Thus, a randomized controlled trial of NMA plots will be conducted. Participants will be randomized to either the rank-heat plot (intervention) or SUCRA plots (control) that present the same NMA results of a study that explored the effectiveness of quality improvement interventions for falls prevention. Outcomes will be ascertained via an online survey. The RCT will take place in an online environment and will require each participant to partake in a single session. This study will help guide best practices for the presentation of reviews to improve the uptake and use of NMA.

ELIGIBILITY:
Inclusion Criteria:

* Clinicians must be accredited to practice in Canada and working (full- or part-time) as a family physician or general internist.

Exclusion Criteria:

* Unable to read and understand English;
* No access to the internet;
* Read, co-authored or peer-reviewed the study: "Quality Improvement strategies to Prevent Falls in the Elderly: A systematic review and network meta-analysis" (manuscript in preparation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who appropriately define the clinical "bottom line." Participants' answers will be independently evaluated by two investigators for agreement with an expert panel's recommendation. | during experiment via single session, <1 hour survey

SECONDARY OUTCOMES:
Proportion of participants who accurately apply the evidence to the provided clinical scenario. | during experiment via single session, <1 hour survey
Completeness of survey data evaluated by two independent investigators | Immediate post-experiment
Time taken to complete survey | Immediate post-experiment